CLINICAL TRIAL: NCT06112873
Title: Development and Validation of Three Mini-questionnaires to Assess the Quality of Life in Food Allergic Patients
Brief Title: Quality of Life in Food Allergy: Validation of Three Mini-questionnaires
Acronym: EVAALIM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University Hospital, Angers (Other Government); University Hospital, Toulouse (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/818
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-06

CONDITIONS: Food Allergy
Keywords: Food Allergy; Quality of Life; Children; Adult; Self-reported questionnaire
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The parents of allergic children 0 to 17 years: The parents of 200 eligible patients will complete the parent questionnaire comprising 15 questions
  Interventions: Other: Quality of Life Questionnaire
- Allergic children aged 8 to 17 years: A total of 200 eligible patients aged 8 to 17 years will complete the children's self-reported questionnaire comprising 13 questions.
  Interventions: Other: Quality of Life Questionnaire
- Adults over 18: A total of 200 adult patients will complete the adult self-reported questionnaire comprising 14 questions.
  Interventions: Other: Quality of Life Questionnaire

INTERVENTIONS:
Other: Quality of Life Questionnaire — Patient (or Parent)-Reported Outcomes via specific questionnaires

SUMMARY:
The evaluation of the quality of life (QOL) in food allergy (AA) is difficult due to the lack of a currently validated questionnaire. There are only a few tools available to assess the impact of nutritional care on the QOL of the allergic patient . Available questionnaires are poorly adapted to studies dealing with large cohorts where functionality and ease of use are determining factors. The aim of this work will be to develop and validate QOL questionnaires for AA, short and easy to use, also integrating the theme of collective catering in order to assess the evolution of QOL in patients with food allergy.

The target population of the questionnaires will be:

i) the parents of allergic children 0 to 17 years (15 questions) ii) allergic children aged 8 to 17 years (13 questions) iii) Adults over 18 (14 questions)

After receiving an information note, eligible patients or their parents will complete the questionnaires. A total of 200 patients will be recruited for each questionnaire.

A statistical evaluation will be carried out using 200 questionnaires for each targeted population in order to validate the psychometric properties of the questionnaire as well as investigate the degree of correlation between the scores of the mini-questionnaire and those obtained using the Europrevall reference questionnaire.

DETAILED DESCRIPTION:
The Réseau d'Allergologie de Franche-Comté (RAFT, University Hospital of Besançon), with the participation of the Allergodiet [1] working group of the French Society of Allergy (SFA), developed this work and contribute to the selection of relevant questions for each age range.

The selected items are divided into three areas: i) social and food limitations; ii) food anxiety; and iii) the risks of accidental ingestion. A statistical evaluation will be carried out using 200 questionnaires for each targeted population in order to validate the psychometric properties of the questionnaire as well as investigate the degree of correlation between the scores of the mini-questionnaire and those obtained using the Europrevall reference questionnaire.

Study Procedures :

After receiving an information note, eligible patients and/or their parents will complete the questionnaires.

Outcome measures:

Patient-Reported Outcomes via specific questionnaires

Participant numbers:

200 patients will be recruited for each questionnaire

Participants and recruitment:

Inclusion criteria :

Patient or parent of a patient with an IgE-mediated allergy to any food, or a non-IgE-mediated allergy to cow's milk in infants.

Exclusion criteria :

All patients who do not fit the inclusion criteria mentioned above, lack of consent, mental or visual disturbances, not understanding the questionnaire language.

Resources :

This multicenter study will be conducted at CHU de Besançon, CHU de Toulouse, CHU Angers and CHU de Lyon.

Data management:

Data will be collected directly from the patients. All paper patient records will be kept in locked filing cabinet. Electronic files will be saved on password protected folder

Oversight :

i) Data will be entered from a professional computer station; ii) all documents containing the identity of the participating subjects (non-objection, list of correspondence, etc.) will be kept away from personal data; iii) if it is a paper document, it will be stored in a secure location known only to professionals involved in the research ; iv) If it is a computerized document, it will be kept on the center's information server with access control by password.

References:

1- Doc, A., Capelli, E., Le Pabic, F., Pouessel, G., Deschildre, A., Morisset, M., & Rame, J. M. (2020). Allergodiet: un groupe de travail de diététiciens nutritionnistes en allergologie. Revue Française d'Allergologie, 60(3), 143-149.

ELIGIBILITY:
Inclusion Criteria:

Patients with an IgE-mediated allergy to any food, or a non-IgE-mediated allergy to cow's milk in infants.

Exclusion Criteria:

All patients who do not fit the inclusion criteria mentioned above, lack of consent, mental or visual disturbances, not understanding the questionnaire language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (or patients parents) cared for food allergy at CHU de Besançon, CHU de Toulouse, CHU Angers and CHU de Lyon including:
  * 200 parents of allergic children
  * 200 allergic children aged 8 to 17 years
  * 200 adults with food allergy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2024-11-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability of Questionnaires | 6 months
Comparability with EUROPREVALL reference questionnaires | 3 months

SECONDARY OUTCOMES:
Discriminative capacity of questionnaires | 3 months

IPD SHARING:
Plan to Share IPD: No